CLINICAL TRIAL: NCT06522009
Title: Effect of Time Delay and Syringe Surface Area on Results of Blood Gas Analysis
Brief Title: Effect of Time Delay and Syringe Surface Area on Blood Gas Samples Analysis
Status: Completed | Type: Observational
Sponsor: Helwan University (Other)
Collaborators: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Adel Ali Hassan, lecturer of anaesthesia, intensive care and pain management, Helwan University
Other Study IDs: 19/4/471
Record Dates: First submitted 2024-07-18; First posted 2024-07-26 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Respiratory Failure
Keywords: blood gas; oxygen saturation; syringe surface area; Time Delay
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To detect the effect of time delay and syringe surface area on the oxygen tension (PaO2), oxyhaemoglobin saturation (SaO2), acidity (pH), and carbon dioxide tension (PaCO2) in both arterial and venous blood gas outcomes.

DETAILED DESCRIPTION:
Arterial blood gas (ABG) analysis and monitoring is a crucial process for the diagnosis and management of the oxygenation status and acid-base balance of high-risk patients during surgery, as well as for the critical care of critically ill patients in the Intensive Care Unit .

Acid-base imbalance anomalies can have major repercussions in a number of medical scenarios, and in a few rare instances, they may even be a risk factor for death.

ABG test explores the arterial blood's pH, oxyhaemoglobin saturation (SaO2), bicarbonate concentration (HCO3), oxygen tension (PaO2), and carbon dioxide tension (PaCO2).

Traditionally, the concept "blood gas testing" has been used to describe measuring the blood's pH, oxygen saturation of haemoglobin (SaO2), and partial pressures of the physiologically active gases (pO2, pCO2). But now available commercial equipment can measure electrolytes (sodium, potassium, chloride, ionized calcium, and magnesium), glucose, lactate, and creatinine, usually all at the same time, in addition to haemoglobin quantification and co-oximetry

ELIGIBILITY:
Inclusion Criteria:

* Critically ill-patients, and intraoperative patients who aged above 18 years.

Exclusion Criteria:

* Patients with haematological diseases e.g. sickle cell anaemia
* burn patients with risk of carbon monoxide poisoning
* ARDS
* pulmonary oedema
* samples that were clotted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill-patients, and intraoperative patients who aged above 18 years.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
To detect the effect of time delay and syringe surface area on the oxygen tension (PaO2) arterial and venous blood gas outcomes. | 1 hour
  PaO2 by mmhg arterial and venous samples
  To detect the effect of time delay and syringe surface area on SO2 in arterial and venous samples
  To detect the effect of time delay and syringe surface area on other parameters of blood gases e.g. PH,CO2

SECONDARY OUTCOMES:
effect of delay on analysis oxyhaemoglobin saturation (SaO2) acidity (pH) carbon dioxide tension (PaCO2) | 60 minutes
  spao2 by mmhg and paco2 by mmhg

CONTACTS AND LOCATIONS:
Overall Officials: Adel A hassan, Md, Principal Investigator — Helwan University
Locations (1):
- Theodor Bilharz Research Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: after the end of the study for one year
Access Criteria: The data will be available upon a reasonable request from the corresponding author.